CLINICAL TRIAL: NCT07313527
Title: PCR for Aspergillus Fumigatus in Blood and Bronchoalveolar Lavage Fluid for Monitoring Cases of Invasive Aspergillosis: What is Its Prognostic Value
Acronym: ASP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9615
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: Invasive Pulmonary Aspergillosis; Aspergillus fumigatus PCR; Bronchoalveolar lavage fluid
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aspergillus fumigatus PCR is currently used in conjunction with serum galactomannan to support the diagnosis of invasive aspergillosis or for monitoring at-risk patients not receiving antifungal prophylaxis. A positive result and a high titer are thought to be associated with the advanced stage of the disease and the fungal load. However, there is limited data on this subject, and no study has primarily focused on the variation of PCR levels during treatment and its potential correlation with treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Positive Aspergillus fumigatus PCR on serum or bronchoalveolar lavage fluid at diagnosis, performed at the Strasbourg University Hospital between January 1, 2017, and December 31, 2024.

Exclusion Criteria:

* No subsequent Aspergillus fumigatus PCR (>24h)
* No diagnosis of probable or proven invasive aspergillosis (EORTC/MSGERC 2020 criteria)
* Effective antifungal treatment against Aspergillus initiated before the first PCR
* Death <72h after starting antifungal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient with positive Aspergillus fumigatus PCR on serum or bronchoalveolar lavage fluid at diagnosis, performed at the Strasbourg University Hospital between January 1, 2017, and December 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Death rate at day 30 in patients with a positive follow-up PCR (blood or bronchoalveolar lavage) | Day 30 post-antifungal treatment
  Death rate at day 30 in patients with a positive follow-up PCR (blood or bronchoalveolar lavage) after the start of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France